CLINICAL TRIAL: NCT01070524
Title: A Randomised, Double-blind, Active-controlled, 3 Way Cross-over Study to Evaluate the Effect on Trough FEV1 After 4 Weeks Treatment With CHF 5188 pMDI qd (Fixed Combination Budesonide / Carmoterol) in Adult Patients With Moderate or Severe Persistent Asthma
Brief Title: Cross-over Study to Evaluate the Effect on Trough Forced Expiratory Volume in One Second (FEV1) After 4 Weeks Treatment With CHF 5188 pMDI qd in Adult Patients With Persistent Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Dr. Dave Singh, The Medicines Evaluation Unit Ltd
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCD-0909-PR-0020; 2009-013759-32 (EudraCT Number)
Record Dates: First submitted 2010-02-17; First posted 2010-02-18 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CHF 5188 pMDI (Experimental)
  Interventions: Drug: CHF 5188 pMDI
- Budesonide extrafine pMDI (Active Comparator)
  Interventions: Drug: Budesonide extrafine pMDI
- Seretide(r) Evohaler(r) (Active Comparator)
  Interventions: Drug: Seretide(r) Evohaler(r)

INTERVENTIONS:
Drug: CHF 5188 pMDI — CHF 5188: fixed combination budesonide/carmoterol
  Arms: CHF 5188 pMDI
Drug: Budesonide extrafine pMDI — Budesonide extrafine pMDI
  Arms: Budesonide extrafine pMDI
Drug: Seretide(r) Evohaler(r) — Seretide(r) Evohaler(r): fixed combination fluticasone/salmeterol
  Arms: Seretide(r) Evohaler(r)

SUMMARY:
Cross-over study to evaluate the effect on trough FEV1 after 4 weeks treatment with CHF5188 pMDI qd in adult patients with persistent asthma

DETAILED DESCRIPTION:
A randomised, double-blind, multinational, multicentre, active-controlled, 3-way cross-over study to evaluate the effect on trough FEV1 after 4 weeks treatment with CHF5188 pMDI qd in adult patients with moderate or severe persistent asthma

ELIGIBILITY:
Inclusion Criteria:

* Moderate or severe asthma partly controlled with ICS or ICS/LABA
* FEV1 ≥ 60% and ≤ 90% of predicted for the patient normal value

Exclusion Criteria:

* Diagnosis of COPD
* History or current evidence of significant cardiovascular disease
* Uncontrolled concomitant disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Trough FEV1 (mean 23h-24h FEV1) | after day 28 dose

SECONDARY OUTCOMES:
Trough FEV1 and forced vital capacity (FVC) (mean 23h-24h) | after day 1 dose
Trough FVC (mean 23-24h) | after day 28 dose
Peak FEV1 and FVC | on day 1 and day 28
FEV1 AUC0-24 | after day 1 and day 28

CONTACTS AND LOCATIONS:
Overall Officials: Dave Singh, MD, Principal Investigator — The Medicines Evaluation Unit Ltd
Locations (1):
- The Medicines Evaluation Unit Ltd, The Langley Building, Southmoor Road, Manchester, United Kingdom

REFERENCES:
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2009-013759-32